CLINICAL TRIAL: NCT01408108
Title: Prospective Randomized Phase III Study of Laparoscopic Lightweight Mesh Repair of Large Hiatal Hernias
Brief Title: Laparoscopic Lightweight Mesh Repair of Large Hiatal Hernias
Acronym: LARGE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odessa National Medical University (Other)
Responsible Party: Principal Investigator, Dr. Andriy V. Malynovskyy, Assistant of department of surgery # 1, Odessa National Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONMU-1
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Hernia, Hiatal
Keywords: Hiatal hernia; Gastro-oesophageal reflux disease; Laparoscopic hiatal repair; Laparoscopic anti-reflux surgery; Partially absorbable lightweight mesh
MeSH Terms: conditions — Hernia, Hiatal; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lightweight mesh repair (Active Comparator): Laparoscopic hiatal repair with sub-lay partially absorbable lightweight mesh
  Interventions: Procedure: Laparoscopic hiatal repair with sub-lay partially absorbable lightweight mesh
- Primary crural repair (Active Comparator): Laparoscopic primary posterior crural repair
  Interventions: Procedure: Laparoscopic primary posterior crural repair

INTERVENTIONS:
Procedure: Laparoscopic hiatal repair with sub-lay partially absorbable lightweight mesh — A fashioned according to the dimensions of hernia defect partially absorbable lightweight mesh Ultrapro™ (Ethicon, Inc.) will be sutured to both crura with 3 to 5 interrupted non-absorbable (Ethibond™ 3-0 by Ethicon, Inc.) sutures (as tension-free repair). Subsequent 2 to 3 interrupted non-absorbable sutures will approximate crura to completely cover a mesh to preclude its contact with the esophagus (original "sandwich" sub-lay technique).
  Other Names: Laparoscopic mesh hiatoplasty; Laparoscopic mesh hiatal closure
  Arms: Lightweight mesh repair
Procedure: Laparoscopic primary posterior crural repair — Posterior cruroraphy will be performed with 3 to 4 interrupted non-absorbable (Ethibond™ 3-0 by Ethicon, Inc.) sutures.
  In the both arms laparoscopic procedure will be done in a standard fashion: reduction of hernia with excision of hernia sac and mobilization of distal esophagus, exposure of borders of hiatal opening including crura posteriorly to esophagus, repair if hiatal hernia defect (30 Fr esophageal bougie is used), a short (2,5 - 3,5 cm) 360° fundoplication wrap (floppy-Nissen procedure) (30 Fr esophageal bougie is used).
  Other Names: Laparoscopic posterior crurorrhaphy; Laparoscopic posterior crural closure
  Arms: Primary crural repair

SUMMARY:
This study is prospective randomized trial enrolling at least 100 participants which compares efficacy and safety of two alternative methods of laparoscopic hiatal repair for large (i.e. with hiatal surface area (HSA) ranging from 10 to 20 sq.cm, which corresponds to diameter of defect from 5 to 8 cm) types I, II, and III hiatal hernias: primary crural repair and repair with partially absorbable lightweight mesh. According to the literature, rates of anatomical failure and recurrence of GERD after primary repair of large hiatal hernias reach 42 %. Mesh repair decreases rates of failures, however, polypropylene and composite PTFE meshes used most widely, result in unacceptable rates of long-term dysphagia and oesophageal strictures. Our own experience of more than 400 repairs using partially absorbable lightweight mesh Ultrapro (Ethicon) and original sub-lay technique of its fixation precluding contact of the mesh with the oesophagus, showed low recurrence rate and a few cases of long-term dysphagia. Thus, final conclusions could be established by prospective randomized study. Our hypothesis is: original technique of lightweight mesh repair is highly effective for prevention of recurrences compared to primary repair and safe in terms of mesh-related dysphagia and oesophageal strictures. The long-term results (24 months post surgery for every patient) will be studied using symptom questionnaires, quality of life and satisfaction questionnaires, barium studies, endoscopic examinations, 24-hour pH testing, and analysis of possible reoperations.

DETAILED DESCRIPTION:
Methods of laparoscopic repair of large and giant hiatal hernias are the most challenging questions in gastrointestinal minimally invasive surgery. The literature demonstrates high rates of anatomical and functional recurrence after laparoscopic repair of large hiatal hernias, particularly following primary crural repair. Different methods of mesh repair were introduced and several trials showed their benefits. However, necessity and method of prosthetic repair remain questionable as mesh repair results in high frequency of long-term dysphagia and oesophageal strictures.

There is insufficient grade 1 evidence for choice of optimal method of repair of large hiatal hernias. Only 3 prospective randomized trials comparing prosthetic and primary hiatal repair were published by Frantzides et al (2002), Granderath et al (2005), and Oelschlager et al (2006). However, these trials could not recommend effective, safe, and relatively inexpensive method of repair. Although Frantzides et al (2002) showed statistically significant decrease of recurrence rate in composite (ePTFE) mesh arm, the study included only patients with diameter of defect 8 cm and greater, thus it is still unknown whether mesh should be used for hernias with smaller diameter of hernia defect, for example, between 5 and 8 cm. Most specialists use mesh when the diameter of the defect is just greater than 5 cm, based on their own experience and widespread literature data, including studies of Champion et al (1998, 2003). In addition, hiatal surface area (HSA), first described by Granderath et al (2007), is more sensitive measure than diameter of hiatal hernia defect, and further trials should focus on it. Finally, ePTFE prosthesis is rather expensive.

The trial of Granderath et al (2005) also was not primarily focused of relation between diameter of hernia defect and rate of recurrences. In this study, recurrence rate was also smaller in the polypropylene arm, but the rate of dysphagia was lager in the same arm. Although later these authors reported that differences between arms in rates of dysphagia and motility disorders vanished in 1 year, most of authors still consider polypropylene mesh potentially unsafe (Frantzides et al, 2010).

To remove the risk of mesh-related oesophageal complications, biological prostheses were introduced for hiatal repair, but the study of Oelschlager et al (2006) demonstrated insignificant difference in recurrence rates in prosthesis arm compared to primary repair arm, although no cases of mesh-related complications were observed in prosthesis arm. Data from the literature and international congresses suggest that biological devices cannot be widely used in the setting of large hiatal hernias due to high rate of recurrences and their high price. Data from another recent numerous publications including reviews made the same conclusions that large and giant hiatal hernias require mesh repair but search for the optimal prosthesis and fashion of its fixation is ongoing.

Hiatal repair by partially absorbable lightweight meshes is promising technique and may become an optimal because it can minimize both recurrences and oesophageal complications. Hazebroek et al (2008) reported good functional, endoscopic, and radiological outcomes in terms of esophageal complications after on-lay placement of titanium-coated lightweight polypropylene mesh (non-randomized prospective study). Our own experience of 400 repairs using lightweight mesh (Ultrapro, Ethicon) and original sub-lay technique of its fixation precluding contact of the mesh with the oesophagus, showed low recurrence rate (4,9%) and a few cases of long-term dysphagia (2,1%). Therefore, the hypothesis of our double-blind prospective randomized trial is: original technique of lightweight mesh (Ultrapro, Ethicon) repair is highly effective for prevention of recurrences compared to primary repair and safe in terms of mesh-related dysphagia and oesophageal strictures.

The study will enroll at least 100 patients with large (i.e. with hiatal surface area (HSA) ranging from 10 to 20 sq.cm, which corresponds to diameter of defect from 5 to 8 cm) types I, II, and III hiatal hernias. The chosen size of the defect is the most questionable in terms of the need for applying a mesh: when HSA is 20 sq.cm or greater the necessity of mesh repair is obvious, when it is less than 10 sq.cm usage of mesh is unreasonable. The basic eligibility criteria will be: absence of oesophageal motility disorders, absence of oesophageal shortening requiring Collis procedure, absence of peptic strictures and other factors that may independently influence the rate of recurrence and dysphagia/oesophageal strictures. Thus, the only difference between arms will be method of hiatal closure. To exclude fundoplication-related bias, standard floppy-Nissen procedure will be performed in every patient.

Every patient will be operated by single surgical team with an experience of more than 1500 laparoscopic anti-reflux procedures since 1998. The necessary ethic regulations will be saved including informed consent with the statement that patient is unaware of the method of repair (double-masked). Every patient is going to be evaluated preoperatively, 6 months, and 24 months postoperatively using symptom questionnaires, quality of life and satisfaction questionnaires, barium studies, endoscopic examinations, and 24-hour pH testing. For issue of efficacy of prosthetic repair, recurrence rate of hernia and GERD, which are the primary outcome measure, will be studied. For issue of safety of prosthetic repair, rates of short- and long-term dysphagia/oesophageal strictures/mesh erosions, which are main secondary outcome measure, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Type I, II and III hiatal hernias, including complicated by GERD
* Able to undergo elective laparoscopic hiatal hernia repair
* Able to 24 months follow-up with office examinations
* Hiatal surface area (HSA) measuring 10 to 20 sq.cm (by granderath et al, 2007) which correspond to the diameter of hernia defect measuring 5 to 8 cm (the distinct size is determined intraoperatively, those with smaller or larger diameter will be excluded from the study)

Exclusion Criteria:

* Unable to undergo laparoscopic hiatal hernia repair due to: severe comorbidities (ASA III and more), previous major surgery with severe adhesions, etc.
* Cases of conversion to open surgery
* Age < 20 years and > 80 years
* BMI < 16 and > 39 kg/m2
* Pregnancy or plans for pregnancy within next 2 years (in females)
* Uncorrectable coagulopathy and immunosuppression
* Oesophageal motility disorders
* Oesophageal peptic strictures
* Oesophageal diverticula, other types (i.e. non-reflux) of chronic esophagitis, connective tissue disorders (e.g. scleroderma)
* Oesophageal shortening (determined intraoperatively as inability to achieve intra-abdominal length of oesophagus at least 3 cm in spite of intramediastinal oesophageal mobilization)
* Barrett's oesophagus
* History of oesophageal/gastric/duodenal surgery including vagotomy
* Relapsing course of ulcer disease/hyperacid gastritis including complicated by delayed gastric/duodenal emptying

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Anatomical and functional recurrence of hiatal hernia and GERD | 24 months
  Recurrence of hiatal hernia, i.e. anatomical recurrence, will be assessed by symptom questionnaire with visual analogue scales, MAINLY by barium study, and data from possible redo procedures. Recurrence of GERD, i.e. functional recurrence, will be evaluated by symptom questionnaire with visual analogue scales, endoscopic examination with assessment of degree of reflux-oesophagitis according to Los-Angeles classification, and 24 hour pH-testing with calculation of DeMeester score.

SECONDARY OUTCOMES:
Repair-related dysphagia/oesophageal stricture/prosthetic erosion | 24 months
  Short- and long-term dysphagia, including due to repair-related oesophageal stricture, will be assessed by symptom questionnaire with visual analogue scales, barium study, endoscopic examination, and data from possible redo procedures. Patients also will be endoscopically assessed for such rare complication as prosthetic erosion of oesophagus.
Quality of life and satisfaction | 24 months
  Quality of life and satisfaction will be assessed by GERD-HRQL score
Operative time | 1 day
Morbidity | 1 month
Postoperative hospital stay | 1 month
Influence on extra-oesophageal complications | 24 months
  Extra-oesophageal complications to be assessed are: asthma, COPD, laryngitis, angina, and arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Volodymyr V. Grubnik, Prof., MD, Principal Investigator — Department of surgery # 1 of Odessa national medical university
Locations (1):
- Department of surgery # 1 of Odessa national medical university, Odessa regional hospital, Odesa, Ukraine

REFERENCES:
- [Background] Frantzides CT, Madan AK, Carlson MA, Stavropoulos GP. A prospective, randomized trial of laparoscopic polytetrafluoroethylene (PTFE) patch repair vs simple cruroplasty for large hiatal hernia. Arch Surg. 2002 Jun;137(6):649-52. doi: 10.1001/archsurg.137.6.649. PMID 12049534
- [Background] Granderath FA, Schweiger UM, Kamolz T, Asche KU, Pointner R. Laparoscopic Nissen fundoplication with prosthetic hiatal closure reduces postoperative intrathoracic wrap herniation: preliminary results of a prospective randomized functional and clinical study. Arch Surg. 2005 Jan;140(1):40-8. doi: 10.1001/archsurg.140.1.40. PMID 15655204
- [Background] Oelschlager BK, Pellegrini CA, Hunter JG, Brunt ML, Soper NJ, Sheppard BC, Polissar NL, Neradilek MB, Mitsumori LM, Rohrmann CA, Swanstrom LL. Biologic prosthesis to prevent recurrence after laparoscopic paraesophageal hernia repair: long-term follow-up from a multicenter, prospective, randomized trial. J Am Coll Surg. 2011 Oct;213(4):461-8. doi: 10.1016/j.jamcollsurg.2011.05.017. Epub 2011 Jun 29. PMID 21715189
- [Background] Champion JK, McKernan JB. Hiatal size and risk of recurrence after laparoscopic fundoplication [abstract]. Surg Endosc. 1998; 12:565-570.
- [Background] Champion JK, Rock D. Laparoscopic mesh cruroplasty for large paraesophageal hernias. Surg Endosc. 2003 Apr;17(4):551-3. doi: 10.1007/s00464-002-8817-7. Epub 2003 Feb 17. PMID 12582773
- [Background] Frantzides CT, Carlson MA, Loizides S, Papafili A, Luu M, Roberts J, Zeni T, Frantzides A. Hiatal hernia repair with mesh: a survey of SAGES members. Surg Endosc. 2010 May;24(5):1017-24. doi: 10.1007/s00464-009-0718-6. Epub 2009 Dec 8. PMID 19997755
- [Background] Hazebroek EJ, Ng A, Yong DH, Berry H, Leibman S, Smith GS. Evaluation of lightweight titanium-coated polypropylene mesh (TiMesh) for laparoscopic repair of large hiatal hernias. Surg Endosc. 2008 Nov;22(11):2428-32. doi: 10.1007/s00464-008-0070-2. Epub 2008 Jul 15. PMID 18626699
- [Background] Granderath FA, Schweiger UM, Pointner R. Laparoscopic antireflux surgery: tailoring the hiatal closure to the size of hiatal surface area. Surg Endosc. 2007 Apr;21(4):542-8. doi: 10.1007/s00464-006-9041-7. Epub 2006 Nov 14. PMID 17103275
- [Background] Grubnik VV, Malynovskyy AV. Laparoscopic repair of hiatal hernias: new classification supported by long-term results. Surg Endosc. 2013 Nov;27(11):4337-46. doi: 10.1007/s00464-013-3069-2. Epub 2013 Jul 23. PMID 23877759